CLINICAL TRIAL: NCT07375953
Title: Repeated Intravenous Thrombolysis for Ischemic Stroke Within 3.0 Hours of Onset With Tenecteplase (RITIS-TNK): a Prospective, Randomized, Open Label, Blinded Assessment of Outcome, and Multi-center Study
Brief Title: Repeated Intravenous Thrombolysis for Ischemic Stroke Within 3.0 Hours of Onset With Tenecteplase (RITIS-TNK)
Acronym: RITIS-TNK
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2025) 501
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental): Tenecteplase is administered intravenously at a dose of 16 mg, with a maximum dose of 0.25 mg/kg.
  Interventions: Drug: Tenecteplase
- Control group (No Intervention): No tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase is administered intravenously at a dose of 16 mg, with a maximum dose of 0.25 mg/kg.
  Arms: TNK group

SUMMARY:
Despite being the standard pharmacological reperfusion therapy for acute ischemic stroke, intravenous thrombolysis is limited by suboptimal recanalization rates. Tenecteplase (TNK), a newer thrombolytic agent, offers practical advantages over alteplase, including single bolus administration. However, a significant proportion of patients fail to achieve early clinical improvement after standard thrombolysis, likely due to persistent vessel occlusion.

This study proposes to investigate a rescue strategy for patients who do not show significant neurological improvement within one hour after receiving standard intravenous tenecteplase within 3 hours of stroke onset. The primary objective is to evaluate the safety and feasibility of administering a second dose of tenecteplase in this scenario. The study will also explore the potential efficacy of this approach in improving recanalization and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year;
* Acute ischemic stroke within 3 hours of onset, having received standard intravenous thrombolysis;
* Measurable neurological deficit before the first intravenous thrombolysis, with NIHSS ≥ 4;
* No significant clinical improvement (reduction in NIHSS ≤ 2) or neurological deterioration after initial improvement at 1 hour after the first thrombolysis, with intracranial hemorrhage ruled out by neuroimaging;
* The second intravenous thrombolysis can be administered within 4.5 hours of onset;
* First stroke onset or past stroke without obvious neurological deficit (mRS≤1);
* Signed informed consent.

Exclusion Criteria:

* Planed for endovascular treatment;
* Significant cerebral white matter hyperintensities (Fazekas score 3)；
* Any coagulation abnormality before the first thrombolysis, including INR > 1.5；
* Pregnancy；
* Allergy to the investigational drug(s)；
* Receipt of dual antiplatelet therapy within 24 hours prior to thrombolysis;
* Comorbidity with other serious diseases;
* Participating in other clinical trials within 3 months;
* Patients not suitable for the study considered by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
proportion of excellent functional outcome (modified Rankin Scale (mRS) 0-1) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
proportion of modified Rankin Scale (mRS) 0-2 | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Scale (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
occurrence of early neurological improvement (ENI) | 24 (-6/+12) hours
  ENI is defined as more than 4-point decrease in National Institute of Health stroke scale score
change in National Institute of Health stroke scale (NIHSS) score | 24 (-6/+12) hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
change in National Institute of Health stroke scale (NIHSS) score | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
new stroke or other vascular event(s) | 90±7 days
symptomatic intracranial hemorrhage (sICH) | 24 (-6/+12) hours
any intracranial hemorrhage | 24 (-6/+12) hours
major systemic bleeding event | 24 (-6/+12) hours
any bleeding event | 24 (-6/+12) hours
all-cause mortality | 90±7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Cui, Shenyang, None Selected, China